CLINICAL TRIAL: NCT00889330
Title: Safety and Efficacy Study of a Eye Drop for Eye Allergy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vistakon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 09-003-05
Record Dates: First submitted 2009-04-24; First posted 2009-04-28 (Estimated); Results first posted 2011-12-08 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-02

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — alcaftadine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- alcaftadine ophthalmic solution (Experimental): active treatment: administered as a single one-drop dose in each eye at each visit (Day 0 and Day 14).
  Interventions: Drug: alcaftadine
- inactive ophthalmic solution vehicle (Placebo Comparator): Placebo, vehicle: administered as a single one-drop dose in each eye at each visit (Day 0 and Day 14).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: alcaftadine — 0.25% Ophthalmic Solution, one drop in each eye at each of two visits.
  Arms: alcaftadine ophthalmic solution
Drug: Placebo — Vehicle without active, one drop in each eye at each of two visits.
  Arms: inactive ophthalmic solution vehicle

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of an anti-allergy eyedrop.

ELIGIBILITY:
Inclusion Criteria:

* At least 10 years of age
* positive history of ocular allergies
* positive skin test reaction to allergens.

Exclusion Criteria:

* known allergy, contraindication, or sensitivities to the use of any of the study medication(s) or their components
* ocular surgical intervention within three (3) months prior to visit 1 or during the study
* known history of retinal detachment, diabetic retinopathy, or progressive retinal disease, or glaucoma
* any other significant illness

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-04; Primary Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Fairfield, Ohio
  - Mason, Ohio

REFERENCES:
- [Derived] Torkildsen G, Shedden A. The safety and efficacy of alcaftadine 0.25% ophthalmic solution for the prevention of itching associated with allergic conjunctivitis. Curr Med Res Opin. 2011 Mar;27(3):623-31. doi: 10.1185/03007995.2010.548797. Epub 2011 Jan 21. PMID 21250860

RESULTS

PARTICIPANT FLOW:
Groups:
- Alcaftadine Ophthalmic Solution: active treatment: administered as a single dose of one drop per eye at each of two visits, Day 0 and Day 14.
- Inactive Vehicle Ophthalmic Solution: inactive treatment: administered as a single dose of one drop per eye at each of two visits, Day 0 and Day 14.
Period: Overall Study
Arm/Group | Alcaftadine Ophthalmic Solution | Inactive Vehicle Ophthalmic Solution
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alcaftadine Ophthalmic Solution | Inactive Vehicle Ophthalmic Solution | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (13.52) | 34.3 (15.64) | 36.1 (40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 15 | 36
  Male | 9 | 15 | 24
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Ocular Itching at Visit 3 (Day 0) at 7 Minutes Following Allergen Challenge, 16 Hours After Treatment Instillation.
Description: A 0 to 4 scale used, allowing for half increment scores, where 0 indicates "none" and 4 indicates "incapacitating itch with an irresistible urge to rub"; measurement taken at up to 7 minutes following allergen challenge, 16 hours post treatment instillation.
Time Frame: Visit 3 (Day 0) 16 hours post-dose, at up to 7 minutes following Allergen Challenge
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alcaftadine Ophthalmic Solution | Inactive Vehicle Ophthalmic Solution
Number analyzed (Participants) | 30 | 30
units on a scale | 0.69 (0.691) | 2.27 (0.970)

2. Primary Outcome: Conjunctival Redness at Visit 3 (Day 0) at 20 Minutes Following Allergen Challenge, 16 Hours After Treatment Instillation
Description: A 0 to 4 scale used, allowing for half increment scores to measure redness, where 0 indicates "none" and 4 indicates "extremely red"; measurement taken at 20 minutes following allergen challenge, 16 hours post treatment instillation.
Time Frame: Visit 3 (Day 0) At 20 minutes following Allergen Challenge, 16 hours post-treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alcaftadine Ophthalmic Solution | Inactive Vehicle Ophthalmic Solution
Number analyzed (Participants) | 30 | 30
units on a scale | 1.96 (0.846) | 2.50 (0.579)

3. Primary Outcome: Ocular Itching at Visit 4 (Day 14) at 7 Minutes Following Allergen Challenge, 15 Minutes Post- Treatment Instillation
Description: 0 to 4 scale, allowing for half increment scores, where 0 indicates "none" and 4 indicates "incapacitating itch with an irresistible urge to rub"
Time Frame: Visit 4 (Day 14) up to 7 minutes following Allergen Challenge
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alcaftadine Ophthalmic Solution | Inactive Vehicle Ophthalmic Solution
Number analyzed (Participants) | 30 | 30
units on a scale | 0.42 (0.509) | 1.90 (1.058)

4. Primary Outcome: Conjunctival Redness at Visit 4 (Day 14) at 20 Minutes Following Allergen Challenge, 15 Minutes Post Treatment Instillation
Description: as for outcome 2
Time Frame: Visit 4 (Day 14) At 20 minutes following Allergen Challenge
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alcaftadine Ophthalmic Solution | Inactive Vehicle Ophthalmic Solution
Number analyzed (Participants) | 30 | 30
units on a scale | 1.57 (0.863) | 2.15 (0.822)

5. Other Pre Specified Outcome: Number of Eyes With a Visual Acuity Change From Visit 1 (Day -21) at Day -14
Description: The number of eyes with any change in visual acuity measurements compared to Day -21.
Time Frame: Visit 2 (Day -14) pre-allergen challenge
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Alcaftadine Ophthalmic Solution | Inactive Vehicle Ophthalmic Solution
Number analyzed (Participants) | 30 | 30
Number analyzed (eyes) | 60 | 60
eyes | 0 | 1

6. Other Pre Specified Outcome: Number of Eyes With a Visual Acuity Change From Visit 1 (Day -21) at Day 0 Pre-dose, Pre-allergen Challenge
Description: The number of eyes with any change in visual acuity measurements compared to Day -21
Time Frame: Visit 3 (Day 0) pre-dose, pre-allergen challenge
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Alcaftadine Ophthalmic Solution | Inactive Vehicle Ophthalmic Solution
Number analyzed (Participants) | 30 | 30
Number analyzed (eyes) | 60 | 60
eyes | 1 | 0

7. Other Pre Specified Outcome: Number of Eyes With a Visual Acuity Change From Visit 1 (Day -21) at Day 14 Pre-dose, Pre-allergen Challenge
Description: The number of eyes with any change in visual acuity measurements compared to Day -21
Time Frame: Visit 4 (Day 14) pre-dose, pre-allergen challenge
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Alcaftadine Ophthalmic Solution | Inactive Vehicle Ophthalmic Solution
Number analyzed (Participants) | 30 | 30
Number analyzed (eyes) | 60 | 60
eyes | 0 | 1

8. Other Pre Specified Outcome: Number of Eyes With a Undilated Fundoscopy Changes From Visit 1 (Day -21) at Day 14
Description: The number of eyes with any change to the following: Vitreous, Retina, Macula, Choroid, Optic Nerve
Time Frame: Visit 4 (Day 14) pre-dose, pre-allergen challenge
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Alcaftadine Ophthalmic Solution | Inactive Vehicle Ophthalmic Solution
Number analyzed (Participants) | 30 | 30
Number analyzed (eyes) | 60 | 60
eyes
  Vitreous | 0 | 0
  Retina | 0 | 0
  Macula | 0 | 0
  Choroid | 0 | 0
  Optic Nerve | 0 | 0

9. Other Pre Specified Outcome: Number of Eyes With Slit Lamp Biomicroscopy Changes From Visit 1 (Day -21) at Day -14
Description: The number of eyes with any change in the following: anterior chamber, conjunctiva, cornea, iris, lens, lids, tear meniscus
Time Frame: Visit 2 (Day -14) pre-allergen challenge
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Alcaftadine Ophthalmic Solution | Inactive Vehicle Ophthalmic Solution
Number analyzed (Participants) | 30 | 30
Number analyzed (eyes) | 60 | 60
eyes
  anterior chamber | 0 | 0
  conjunctiva | 0 | 0
  cornea | 0 | 0
  iris | 0 | 0
  lens | 0 | 0
  lids | 0 | 0
  tear meniscus | 0 | 0

10. Other Pre Specified Outcome: Number of Eyes With Slit Lamp Biomicroscopy Changes From Visit 1 (Day -21) at Day 0 Pre-dose, Pre-allergen Challenge
Description: as for outcome 9
Time Frame: Visit 3 (Day 0) pre-dose, pre-allergen challenge
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Alcaftadine Ophthalmic Solution | Inactive Vehicle Ophthalmic Solution
Number analyzed (Participants) | 30 | 30
Number analyzed (eyes) | 60 | 60
eyes
  anterior chamber | 0 | 0
  conjunctiva | 0 | 0
  cornea | 0 | 0
  iris | 0 | 0
  lens | 0 | 0
  lids | 1 | 0
  tear meniscus | 0 | 0

11. Other Pre Specified Outcome: Number of Eyes With Slit Lamp Biomicroscopy Changes From Visit 1 (Day -21) at Day 0 Post-dose, Pre-allergen Challenge
Description: as for outcome 9
Time Frame: Visit 3 (Day 0) post-dose, pre-allergen challenge
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Alcaftadine Ophthalmic Solution | Inactive Vehicle Ophthalmic Solution
Number analyzed (Participants) | 30 | 30
Number analyzed (eyes) | 60 | 60
eyes
  anterior chamber | 0 | 0
  conjunctiva | 0 | 0
  cornea | 0 | 0
  iris | 0 | 0
  lens | 0 | 0
  lids | 1 | 0
  tear meniscus | 0 | 0

12. Other Pre Specified Outcome: Number of Eyes With Slit Lamp Biomicroscopy Changes From Visit 1 (Day -21) at Day 14 Pre-dose, Pre-allergen Challenge
Description: as for outcome 9
Time Frame: Visit 4 (Day 14) pre-dose, pre-allergen challenge
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Alcaftadine Ophthalmic Solution | Inactive Vehicle Ophthalmic Solution
Number analyzed (Participants) | 30 | 30
Number analyzed (eyes) | 60 | 60
eyes
  anterior chamber | 0 | 0
  conjunctiva | 0 | 0
  cornea | 0 | 0
  iris | 0 | 0
  lens | 0 | 0
  lids | 1 | 0
  tear meniscus | 0 | 0

13. Other Pre Specified Outcome: Number of Eyes With Slit Lamp Biomicroscopy Changes From Visit 1 (Day -21) at Day 14 Post-dose, Pre-allergen Challenge
Description: as for outcome 9
Time Frame: Visit 4 (Day 14) post-dose, pre-allergen challenge
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Alcaftadine Ophthalmic Solution | Inactive Vehicle Ophthalmic Solution
Number analyzed (Participants) | 30 | 30
Number analyzed (eyes) | 60 | 60
eyes
  anterior chamber | 0 | 0
  conjunctiva | 0 | 0
  cornea | 0 | 0
  iris | 0 | 0
  lens | 0 | 0
  lids | 1 | 0
  tear meniscus | 0 | 0

ADVERSE EVENTS:
Arm/Group | Alcaftadine Ophthalmic Solution | Inactive Vehicle Ophthalmic Solution
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other